CLINICAL TRIAL: NCT02086240
Title: Reproducibility of the 11C-PBR28 PET Signal
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects recruited
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13HH1842
Record Dates: First submitted 2014-02-11; First posted 2014-03-13 (Estimated); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Neurodegenerative Disorders
MeSH Terms: conditions — Neurodegenerative Diseases | interventions — N-benzyl-N-ethyl-2-(7,8-dihydro-7-methyl-8-oxo-2-phenyl-9H-purin-9-yl)acetamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- XBD173 (Experimental): XBD173 (Emapunil is an anxiolytic drug which acts as a selective agonist at the peripheral benzodiazepine receptor), a drug which binds the TSPO with high affinity. In a previous study (approved by NRES Committee London-West London, REC ref No. 12/LO/0735), we administered an oral dose of XBD173 (up to 90mg) in 12 subjects. No adverse events due to XBD173 occurred and it was well tolerated.
  Interventions: Drug: XBD173

INTERVENTIONS:
Drug: XBD173 — XBD173 (Emapunil is an anxiolytic drug which acts as a selective agonist at the peripheral benzodiazepine receptor), a drug which binds the TSPO with high affinity.
  Other Names: Emapunil

SUMMARY:
The Translocator Protein (TSPO) is a protein which reaches very high levels when there is inflammation in the brain.

Recently, radioligands have been developed which attach to the TSPO (a radioligand is a drug which has been tagged with radioactivity). Using positron emission tomography (PET) imaging, the radioligand can be detected following injection into a patient. However, it is difficult to accurately measure the amount of TSPO using PET at the moment. This is because the brain does not have a "reference region" for TSPO (ie an area in the brain with no TSPO at all). "Reference regions" are very useful to help work out how much of a PET signal represents "specific binding" (of the radioligand to the target of interest), and how much represents "non specific binding" (of the radioligand to many other structures which are not of interest). In the absence of a reference region, non specific binding can be estimated by giving a drug which binds to the TSPO.

The drug prevents the radioligand binding the TSPO and (in a manner of speaking) "creates" a temporary reference region so non specific binding can be measured. To do this, we will use XBD173 (Emapunil is an anxiolytic drug which acts as a selective agonist at the peripheral benzodiazepine receptor) to bind TSPO and block binding of the PET ligand ([11C]PBR28), a TSPO ligand from the phenoxyarlyacetamide class.

Most TSPO PET studies (and in one of our previous studies approved by West London REC) quantify the signal using a ratio of specific binding in the brain to radioactivity in the blood. This requires arterial line insertion which is burdensome for subjects, and increases variability. In this study we aim to determine the ratio of specific binding in the brain to nonspecific binding in the brain by using the temporary reference region. For more accuracy the participants will repeat the scanning procedure so determine test-retest variability of the amount of TSPO.

DETAILED DESCRIPTION:
The Translocator Protein (TSPO) is a protein which reaches very high levels when there is inflammation in the brain.

Recently, radioligands have been developed which attach to the TSPO (a radioligand is a drug which has been tagged with radioactivity). Using positron emission tomography (PET) imaging, the radioligand can be detected following injection into a patient. However, it is difficult to accurately measure the amount of TSPO using PET at the moment. This is because the brain does not have a "reference region" for TSPO (ie an area in the brain with no TSPO at all). "Reference regions" are very useful to help work out how much of a PET signal represents "specific binding" (of the radioligand to the target of interest), and how much represents "non specific binding" (of the radioligand to many other structures which are not of interest). In the absence of a reference region, non specific binding can be estimated by giving a drug which binds to the TSPO.

The drug prevents the radioligand binding the TSPO and (in a manner of speaking) "creates" a temporary reference region so non specific binding can be measured. The aim of this study, therefore, is to develop a method to allow accurate quantification of TSPO expression in the brain of healthy subjects. The study will also include patients with multiple sclerosis to determine the reproducibility of the 11C-PBR28 PET signal in a population which is characterised by a raised TSPO signal. This is vital since 11C-PBR28 PET signal is being evaluated as a marker of disease activity and treatment response, in conditions characterised by neuroinflammation including MS. If there is high test re-test variability in people with raised TSPO signal, this argues against the usefulness of 11C-PBR28 PET for these purposes.To do this, we will use XBD173 (Emapunil is an anxiolytic drug which acts as a selective agonist at the peripheral benzodiazepine receptor) to bind TSPO and block binding of the PET ligand ([11C]PBR28), a TSPO ligand from the phenoxyarlyacetamide class. Because different people possess different types of TSPO (due to a genetic difference between subjects, there are 3 types of TSPO expression patterns) it will be important to study subjects from each of the 3 groups.

We will study healthy volunteers and patients with multiple sclerosis. Each subject will undergo:

1. Screening visit, to take blood and determine the TSPO subtype of the subject.
2. Study day 1: the subject will undergo two PET/CT scans and an MRI scan of the brain. This will involve insertion of an arterial line. In between the two PET scans, the subject will be given an oral dose of XBD173 (up to 90mg).
3. Study day 2: Repeat of the procedures of Study day 1. Only one MRI scan will be done during one of the two study visits. Recruitment Healthy volunteers will be recruited from posters (including e-posters on electronic notice boards and emails), announcements in lectures, and word of mouth around Imperial College campuses. MS patients will be recruited from Neurology clinics across the Imperial Healthcare NHS Trust Hospitals, such as Charing Cross Hospital and St Mary's Hospital. Patients may be referred from University College London Hospital and National Hospital for Neurology and Neurosurgery if suitable for the study.

Male or female participants between 18 to 70 will be included. Women of child bearing potential will undergo a urinary pregnancy test prior to scanning to ensure they are not pregnant.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 70 years of age inclusive, at the time of signing the informed consent.
2. Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, and laboratory tests.
3. A female subject is eligible to participate if she is a) of non-childbearing potential, defined as premenopausal females with a documented tubal ligation or hysterectomy, or postmenopausal defined as 12 months of spontaneous amenorrhea or b) of childbearing potential but not pregnant (as determined by urinary pregnancy test on screening and on each study day) and willing to use one of the contraception methods listed below.
4. Male subject must agree to use one of the contraception methods listed below.
5. Able to lie comfortably on back for up to 90 minutes at a time.
6. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

1. Any clinical significant medical conditions that in the opinion of the investigator would compromise subjects' safety or compliance with study procedures.
2. Any clinical condition which in the opinion of the principal investigator would compromise the scientific integrity of the study.
3. Unwillingness or inability to follow the procedures outlined in the protocol.
4. Subject is mentally or legally incapacitated.
5. Presence of a cardiac pacemaker or other electronic device or ferromagnetic metal foreign bodies as assessed by a standard pre-MRI questionnaire.
6. Contraindications to blood sampling and arterial cannulation.
7. Positive Allen's test.
8. Prolonged Prothrombin Time.
9. Participation in a research study involving ionisation radiation within the last 3 years.
10. Significant radiation exposure other than dental Xrays in last 1 year.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2018-01 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
TSPO Binding Status | Baseline/Screening visit
  Participants will be screened to determine TSPO genotype at the rs6971 polymorphism from a venous blood sample.

OTHER OUTCOMES:
To determine test re-test variability of both BPND and VT for [11C]PBR28 in healthy volunteers and MS patients. | 1st and 2nd Study Visit (approximately 10 days after the 1st study visit)
  Determination of test re-test variability of both BPND and VT for 11CPBR28 in healthy volunteers and MS patients. Subjects will receive a baseline 11C-PBR28 scan, and then a repeat scan following an oral dose of 90mg XBD173 (Emapunil). Both VT and BPND will be determined. Subjects will then return approximately 10 days later for a repeat of these procedures.

CONTACTS AND LOCATIONS:
Overall Officials: David Owen, PhD, Principal Investigator — Imperial College London
Locations (1):
- NIHR/Wellcome Trust Imperial Clinical Research Facility, London, United Kingdom